CLINICAL TRIAL: NCT05395832
Title: Effectiveness of Two Video-based Multicomponent Treatments for Fibromyalgia: The Added Value of Face-to-face Sesions in Nature or at Sea in a Three-arm Randomised Controlled Trial
Brief Title: Effectiveness of Video-based Multicomponent Treatment for Fibromyalgia Plus Face-to-face Sesions in Nature or at Sea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Universitat Autonoma de Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FIBROWALK NATURE
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; multicomponent treatment; chronic pain; pain neuroscience education; therapeutic exercise; cognitive behavioural therapy; mindfulness; randomized controlled trial; virtual format
MeSH Terms: conditions — Fibromyalgia; Chronic Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TAU + multicomponent treatment VIRTUAL FIBROWALK at sea (Experimental): VIRTUAL FIBROWALK is a multicomponent non-pharmacological program based on Pain Neuroscience Education (PNE), therapeutic exercise, Cognitive Behavioural Therapy (CBT) and Mindfulness Training. In this arm a 4 face-to-face session at sea will be added to solve doubts and emphasize the most important points of therapy
  Interventions: Behavioral: TAU + multicomponent treatment VIRTUAL FIBROWALK + 4 face-to-face sessions at sea
- TAU + multicomponent treatment VIRTUAL FIBROWALK in nature (Active Comparator): VIRTUAL FIBROWALK is a multicomponent non-pharmacological program based on Pain Neuroscience Education (PNE), therapeutic exercise, Cognitive Behavioural Therapy (CBT) and Mindfulness Training. In this arm a 4 face-to-face session in nature will be added to solve doubts and emphasize the most important points of therapy
  Interventions: Behavioral: TAU + multicomponent treatment VIRTUAL FIBROWALK + 4 face-to-face sessions in nature
- TAU + multicomponent treatment VIRTUAL FIBROWALK (Active Comparator): VIRTUAL FIBROWALK is a multicomponent non-pharmacological program based on Pain Neuroscience Education (PNE), therapeutic exercise, Cognitive Behavioural Therapy (CBT) and Mindfulness Training
  Interventions: Behavioral: TAU + multicomponent treatment VIRTUAL FIBROWALK

INTERVENTIONS:
Behavioral: TAU + multicomponent treatment VIRTUAL FIBROWALK + 4 face-to-face sessions at sea — Group treatment protocol of 12 weekly 60 minute virtual sessions. All sessions include the following ingredients (approx. in the same order):
  Pain neuroscience education (15 min.) Cognitive restructuring (15 min.) Mindfulness techniques (15 min.) Physical exercise(15 min.) Treatment as Usual (TAU) 4 face-to-face sessions (1 per mounth) at sea Standard pharmacological treatment usually provided to patients with fibromyalgia.
  Arms: TAU + multicomponent treatment VIRTUAL FIBROWALK at sea
Behavioral: TAU + multicomponent treatment VIRTUAL FIBROWALK + 4 face-to-face sessions in nature — Group treatment protocol of 12 weekly 60 minute virtual sessions. All sessions include the following ingredients (approx. in the same order):
  Pain neuroscience education (15 min.) Cognitive restructuring (15 min.) Mindfulness techniques (15 min.) Physical exercise(15 min.) Treatment as Usual (TAU) 4 face-to-face sessions (1 per mounth) in nature Standard pharmacological treatment usually provided to patients with fibromyalgia.
  Arms: TAU + multicomponent treatment VIRTUAL FIBROWALK in nature
Behavioral: TAU + multicomponent treatment VIRTUAL FIBROWALK — Group treatment protocol of 12 weekly 60 minute virtual sessions. All sessions include the following ingredients (approx. in the same order):
  Pain neuroscience education (15 min.) Cognitive restructuring (15 min.) Mindfulness techniques (15 min.) Physical exercise(15 min.) Treatment as Usual (TAU) Standard pharmacological treatment usually provided to patients with fibromyalgia.
  Arms: TAU + multicomponent treatment VIRTUAL FIBROWALK

SUMMARY:
The aim of this study was to examine the effectiveness of a video-based multicomponent program: the Fibrowalk Virtual plus face-to-face sessions for patients with fibromyalgia (FM) in nature or at sea (FM) compared to Fibrowalk Virtual only.

DETAILED DESCRIPTION:
This is a tree-arm RCT focused on the safety and potential effectiveness of the multicomponent program VIRTUAL FIBROWALK as coadjuvant of treatment-as- usual (TAU) in comparation of the Fibrowalk virtual plus face-to-face sessions in the nature or at sea.

VIRTUAL FIBROWALK combines multicomponent approach based on Pain Neuroscience Education (PNE), therapeutic exercise, Cognitive Behavioural Therapy (CBT) and Mindfulness training.

FACE-TO-FACE SESSIONS ADDED TO VIRTUAL FIBROWALK combines de same components than Fibrowalk Virtual and added 4 face-to-face sessions (1 per mounth) to resolve doubts and reinforce the main concepts of therapy in the nature or at sea.

The main hypothesis is that improvement on functional impairment of patients with fibromyalgia can be achieved by the direct intervention on mechanisms such as kinesiophobia and fear avoidance

ELIGIBILITY:
Inclusion Criteria:

* Adults from 18 to 75 years-old. 1990 American College of Rheumatology (ACR) classification criteria + the 2011 modified - - - ACR diagnostic criteria for fibromyalgia
* Able to understand Spanish and accept to participate in the study.

Exclusion Criteria:

* Participating in concurrent or past RCTs (previous year).
* Comorbidity with severe mental disorders (i.e. psychosis) or neurodegenerative diseases (i.e. Alzheimer) that that would limit the ability of the patient to participate in the RCT.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2022-09-25 (Estimated); Study Completion 2023-02-23 (Estimated)

PRIMARY OUTCOMES:
Revised Fibromyalgia Impact Questionnaire (FIQR) | Through study completion, an average of 3 months
  The FIQR comprises three dimensions: physical dysfunction (scores from 0 to 30), overall impact (scores from 0 to 20), and intensity of the symptoms (scores from 0 to 50) is used to measure the impact generated by FM during the last week. It consists of 21 items, which are answered on a numerical rating scale of 11 points (from 0 to 10). Total scores can range from 0 to 100, with higher scores reflecting greater deterioration.

SECONDARY OUTCOMES:
Visual-analogue scale of perceived pain (VAS-Pain) | Through study completion, an average of 3 months
  Patients indicate their pain during the last week on a 10 cm line. Total scores range from 0 to 10, where higher scores indicate a greater pain.
Tampa Scale for Kinesiophobia (TSK-11) | Through study completion, an average of 3 months
  TSK-11 is used to assess fear of pain and movement. It consists of 11 items, which are answered on a Likert scale of 4 points. Total scores of each scale range from 11 to 44, where higher scores indicate a greater fear of pain and movement.
Hospital Anxiety and Depression Scale (HADS) | Through study completion, an average of 3 months
  HADS is used to quantify the severity of anxiety and depression symptoms. It consists of two dimensions (anxiety and depression) of 7 items each responding on a Likert scale of 4 points. Total scores of each scale (HADS-A and HADSD) range from 0 to 21, where higher scores indicate greater severity of symptoms.
Physical Function of the 36-Item Short Form Survey (SF-36) | Through study completion, an average of 3 months
  Physical Function of the 36-Item Short Form Survey (SF-36) was used to measure physical function.This dimension comprises a total of 10 items, which are answered on a Likert scale of 3 points. Total scores on each scale are then transformed and can range from 0 to 100, with higher scores indicate better physical function.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Vall Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No